NCT number: NCT05683158

## Research protocol (Human subject study)

## Research project title

Compensatory kinematic analysis in various directions after chronic stroke

## Methodology and Design

The inclusion criteria for the participants with stroke were physician-confirmed chronic hemiplegia ( $\geq$  6 months onset), Mini-Mental State Examination  $\geq$  25, Modified Ashworth Scale (MAS) (biceps  $\leq$  2, triceps  $\leq$  2), ability to sit alone on a chair, and FMA upper extremities score  $\geq$  21. The healthy participants were individuals without any history of neurological or orthopedic diseases.

- The exclusion criteria were muscle flaccidity, neglect syndrome, orthopaedic diseases, and poor coordination.
- \* The specific placement of markers



- Sternum, xyphoid process, Both acromion, C7, T4, elbow(lateral and medial epicondyle), wrist (lateral and medial styloid process), finger 3<sup>rd</sup> MCP

The seated reaching task posture is as follows:





- The participant attempts to reach the target using the affected upper limb
- The seated height is adjusted to 100% of the participant's lower limb length, with the feet flat on the floor and the knees bent at a 90 degree angle. A chair with adjustable height is used to achieve this.
- Reaching movements are categorized into three directions: forward, ipsilateral and contralateral direction.
- The task is performed five times in a comfortable speed for each direction, and for analysis purposes, three out of the five trials are selected to calculate the average time.

#### 1. Clinical assessment

# 1-1. Fugl-Meyer motor Assessment of the Lower Extremity (FMA-UE) Assessment of sensorimotor function:

| | $\mathbf{Y}$ , sitting po | sition | | | | |
|---|---|---|---|---|---|---|
| I. Reflex activity | | | none | can be e | elicited | |
| Flexors: biceps and finger flexors (at least one) | | | 0 | 2 | | |
| Extensors: triceps | • | , | | 0 2 | | |
| | | | Subtotal I (max | 4) | | |
| II. Volitional moveme | nt within s | svneraies. | without gravitational help | none | partial | full |
| Flexor syneray: Hand from | | Shoulder | retraction | 0 | 1 | 2 |
| contralateral knee to ipsilate | | Silouidei | elevation | 0 | 1 1 | 2 |
| From extensor synergy (she | oulder | | abduction (90°) | Ö | 1 1 | 2 |
| adduction/internal rotation, | | | external rotation | ő | 1 | 2 |
| extension, forearm pronation | | Elbow | flexion | ő | i | 2 |
| synergy (shoulder abductio | | Forearm | supination | 0 | i | 2 |
| rotation, elbow flexion, fore | arm | | | | | |
| supination). | | Shoulder | adduction/internal rotation | 0 | 1 | 2 |
| Extensor synergy: Hand f | | Elbow | extension | 0 | 1 | 2 |
| ipsilateral ear to the contral | ateral knee | Forearm | pronation | 0 | 1 | 2 |
| | | 4.5.5 | Subtotal II (max 1 | 3) | | |
| III. Volitional moveme | | | | none | partial | full |
| Hand to lumbar spine | | | in front of ant-sup iliac spine | 0 | | |
| hand on lap | | | c spine (without compensatior | 1) | 1 | |
| ** | | | ithout compensation) | | | 2 |
| Shoulder flexion 0°- 90° | | | elbow flexion | 0 | | |
| elbow at 0° | | | on during movement | | 1 | |
| pronation-supination 0° | | | abduction or elbow flexion | | | 2 |
| Pronation-supination | | | starting position impossible | 0 | | |
| elbow at 90° | limited pronation/supination, maintains starting position | | CIT | | | |
| houlder at 0° full pronation/supination, maintains starting position | | | | 2 | | |
| COLLD | | | Subtotal III (max | 3) | | |
| IV. Volitional movement with little or no synergy | | none | partial | full | | |
| Shoulder abduction 0 - 90 | )° immedia | ate supination | or elbow flexion | 0 | | |
| elbow at 0° | supination | tion or elbow flexion during movement | | | 1 | |
| forearm neutral | | | ains extension and pronation | | | 2 |
| Shoulder flexion 90° - 180° immediate abduction or elbow flexion | | 0 | | | | |
| | | | exion during movement | | 1 | |
| pronation-supination 0° | | flexion 180°, no shoulder abduction or elbow flexion | | | | 2 |
| Pronation/supination | | | on, starting position impossibl | | | |
| elbow at 0° | | | ination, maintains start positio | | 1 | 77.00 |
| shoulder at 30°- 90° flexion | | | | 2 | | |
| Subtotal IV (max 6) | | | 3) | | | |
| V. Normal reflex active part IV; compare with the u | | | score of 6 points is achieved in | hyper | lively | normal |
| 2 | | | peractive | 0 | | |
| Biceps, triceps, | | 3 reflexes markedly hyperactive effex markedly hyperactive or at least 2 reflexes lively | | " | 1 | |
| | ximum of 1 reflex lively, none hyperactive | | | | 2 | |
| finger flexors | maximum of 1 reflex lively, none hyperactive Subtotal V (max 2) | | | | | |
| finger flexors m | aximum or r | | Subtotal V (max : | 2) | | |
| finger flexors m | aximum or 1 | • | Subtotal V (max | 2) | | |



| B. WRIST support may be provided at the elbow to take or hold the starting | | | partial | full |
|---|---|---|---|---|
| position, no support at wrist, check the passive range of motion prior testing | | | <b>J</b> | 1 4111 |
| Stability at 15° dorsiflexion | less than 15° active dorsiflexion | 0 | | |
| elbow at 90°, forearm pronated | dorsiflexion 15°, no resistance tolerated | | 1 | |
| shoulder at 0° | maintains dorsiflexion against resistance | | | 2 |
| Repeated dorsifexion / volar flexion | cannot perform volitionally | 0 | | |
| elbow at 90°, forearm pronated | limited active range of motion | | 1 | |
| shoulder at 0°, slight finger flexion | full active range of motion, smoothly | | | 2 |
| Stability at 15° dorsiflexion | less than 15° active dorsiflexion | 0 | | |
| elbow at 0°, forearm pronated | dorsiflexion 15°, no resistance tolerated | | 1 | l |
| slight shoulder flexion/abduction | maintains dorsiflexion against resistance | | | 2 |
| Repeated dorsifexion / volar flexion cannot perform volitionally | | 0 | | |
| elbow at 0°, forearm pronated | limited active range of motion | | 1 | |
| slight shoulder flexion/abduction | full active range of motion, smoothly | | | 2 |
| Circumduction | cannot perform volitionally | 0 | | |
| elbow at 90°, forearm pronated | jerky movement or incomplete | | 1 | l |
| shoulder at 0° | complete and smooth circumduction | | | 2 |
| | Total B (max 10) | | | |

| <b>C. HAND</b> support may be provided at the elbow to keep 90° flexion, no support at the wrist, compare with unaffected hand, the objects are interposed, active grasp | | | partial | full |
|---|---|---|---|---|
| Mass flexion | | 0 | 1 | 2 |
| from full active or passive extension | | | | |
| Mass extension | G + GOTH | 0 | 1 | 2 |
| from full active or passive flexion | (A) (S) | U | 1 | |
| GRASP | | | | |
| a. Hook grasp | cannot be performed | 0 | | |
| flexion in PIP and DIP (digits II-V), | can hold position but weak | | 1 | |
| extension in MCP II-V | maintains position against resistance | | | 2 |
| b. Thumb adduction | cannot be performed | 0 | | |
| 1-st CMC, MCP, IP at 0°, scrap of paper | can hold paper but not against tug | | 1 | |
| between thumb and 2-nd MCP joint | can hold paper against a tug | | | 2 |
| c. Pincer grasp, opposition | cannot be performed | 0 | | |
| pulpa of the thumb against the pulpa of | can hold pencil but not against tug | | 1 | |
| 2-nd finger, pencil, tug upward | can hold pencil against a tug | CI | | 2 |
| d. Cylinder grasp | cannot be performed | 0 | | 1 |
| cylinder shaped object (small can) | can hold cylinder but not against tug | | 1 | |
| tug upward, opposition of thumb and | can hold cylinder against a tug | | | 2 |
| fingers | | | | |
| e. Spherical grasp | cannot be performed | 0 | | ) · |
| fingers in abduction/flexion, thumb | can hold ball but not against tug | 1000 | 1 | |
| opposed, tennis ball, tug away | can hold ball against a tug | | | 2 |
| | Total C (max 14) | | | |

| D. COORDINATION closed, tip of the index f | marked | slight | none | |
|---|---|---|---|---|
| Tremor | | 0 | 1 | 2 |
| Dysmetria | pronounced or unsystematic<br>slight and systematic<br>no dysmetria | 0 | 1 | 2 |
| | | ≥ 6s | 2 - 5s | < 2s |
| Time<br>start and end with the<br>hand on the knee | 6 or more seconds slower than unaffected side<br>2-5 seconds slower than unaffected side<br>less than 2 seconds difference | 0 | 1 | 2 |
| | Total D (max 6) | | | |



## 1-2 TIS

| Item | Item | | |
|---|---|---|---|
| 1 | Static sitting balance<br>Starting position | Patient falls or cannot maintain starting position for 10 seconds without arm support Patient can maintain starting position for 10 seconds If score = 0, then TIS total score = 0 | □ 0<br>□ 2 |
| 2 | Starting position<br>Therapist crosses the unaffected leg over the hemiplegic leg | Patient falls or cannot maintain sitting position for 10 seconds without arm support Patient can maintain sitting position for 10 seconds | □ 0<br>□ 2 |
| 3 | Starting position Patient crosses the unaffected leg over the hemiplegic leg | Patient falls Patient cannot cross the legs without arm support on bed or table Patient crosses the legs but displaces the trunk more than 10 cm backwards or assists crossing with the hand Patient crosses the legs without trunk displacement or assistance Total static sitting balance | □ 0<br>□ 1<br>□ 2<br>□ 3<br>/7 |
| 1 | Dynamic sitting balance Starting position Patient is instructed to touch the bed or table with the hemiplegic elbow (by shortening the hemiplegic side and lengthening the unaffected side) and return to the starting position | Patient falls, needs support from an upper extremity or the elbow does not touch the bed or table Patient moves actively without help, elbow touches bed or table If score = 0, then items 2 and 3 score 0 | □ 0<br>□ 1 |
| 2 | Repeat item 1 | Patient demonstrates no or opposite shortening/lengthening Patient demonstrates appropriate shortening/lengthening If score = 0, then item 3 scores 0 | □ 0<br>□ 1 |
| 3 | Repeat item 1 | Patient compensates. Possible compensations are: (1) use of upper extremity, (2) contralateral hip abduction, (3) hip flexion (if elbow touches bed or table further then proximal half of femur), (4) knee flexion, (5) sliding of the feet Patient moves without compensation | □ 0<br>□ 1 |
| 4 | Starting position Patient is instructed to touch the bed or table with the unaffected elbow (by shortening the unaffected side and lengthening the hemiplegic side) and return to the starting position | Patient falls, needs support from an upper extremity or the elbow does not touch the bed or table Patient moves actively without help, elbow touches bed or table If score = 0, then items 5 and 6 score 0 | □ 0<br>□ 1 |
| 5 | Repeat item 4 | Patient demonstrates no or opposite shortening/lengthening Patient demonstrates appropriate shortening/lengthening If score = 0, then item 6 scores 0 | □ 0<br>□ 1 |

| Patient compensates. Possible compensations are: (1) use of upper certremity, (2) contralateral hip abduction, (3) hip flexion (if elbow touches bed or table further then proximal half of femur), (4) knee flexion, (5) sliding of the feet Patient moves without compensation 1 | Item | | | |
|---|---|---|---|---|
| Patient is instructed to lift pelvis from bed or table at the hemiplegic side (by shortening the hemiplegic side and lengthening the unaffected side) and return to the starting position Repeat item 7 Patient compensates. Possible compensations are: (1) use of upper extremity, (2) pushing off with the ipsilateral foot (heel loses contact with the floor) Patient is instructed to lift pelvis from bed or table at the unaffected side phening the hemiplegic side) and return to the starting position Patient is instructed to lift pelvis from bed or table at the unaffected side (by shortening the unaffected side and lengthening the hemiplegic side) and return to the starting position Repeat item 9 Patient compensates. Possible compensations are: (1) use of upper extremity, (2) pushing off with the ipsilateral foot (heel loses contact with the floor) Patient demonstrates appropriate shortening/lengthening If score = 0, then item 10 scores 0 Patient compensates. Possible compensations are: (1) use of upper extremities, (2) pushing off with the ipsilateral foot (heel loses contact with the floor) Patient moves without compensation are: (1) use of upper extremities, (2) pushing off with the ipsilateral foot (heel loses contact with the floor) Patient moves without compensation Total dynamic sitting balance Co-ordination 1 Starting position Patient is instructed to rotate upper trunk 6 times (every shoulder should be moved forward 3 times), first side that moves must be hemiplegic side, head should be fixated in starting position Patient is instructed to rotate lower trunk 6 times (every knee should be moved forward 3 times), first side that moves must be hemiplegic side, upper trunk should be fixated in starting position Patient is instructed to rotate lower trunk 6 times (every knee should be moved forward 3 times), first side that moves must be hemiplegic side, upper trunk should be fixated in starting position Patient is instructed to rotate lower trunk 6 times (every knee should be moved forward 3 times), first | 6 | Repeat item 4 | extremity, (2) contralateral hip abduction, (3) hip flexion (if elbow touches bed or table further then proximal half of femur), (4) knee flexion, (5) sliding of the feet | |
| extremity, (2) pushing off with the ipsilateral foot (heel loses contact with the floor) Patient moves without compensation | 7 | Patient is instructed to lift pelvis from bed or table at the hemiplegic side (by shortening the hemiplegic side and lengthening | shortening/lengthening Patient demonstrates appropriate shortening/lengthening | |
| Patient is instructed to lift pelvis from bed or table at the unaffected side (by shortening the unaffected side and lengthening the hemiplegic side) and return to the starting position Repeat item 9 Patient compensates. Possible compensations are: (1) use of upper extremities, (2) pushing off with the ipsilateral foot (heel loses contact with the floor) Patient moves without compensation Patient is instructed to rotate upper trunk 6 times (every shoulder should be moved forward 3 times), first side that moves must be hemiplegic side, head should be fixated in starting position Repeat item 1 within 6 seconds Rotation is asymmetrical Rotation is asymmetrical Starting position Patient is instructed to rotate lower trunk 6 times (every knee should be moved forward 3 times), first side that moves must be hemiplegic side, head should be fixated in starting position Rotation is asymmetrical Starting position Patient is instructed to rotate lower trunk 6 times (every knee should be moved forward 3 times), first side that moves must be hemiplegic side, upper trunk should be fixated in starting position Repeat item 3 within 6 seconds Rotation is asymmetrical | 8 | Repeat item 7 | extremity, (2) pushing off with the ipsilateral foot (heel loses contact with the floor) | |
| extremities, (2) pushing off with the ipsilateral foot (heel loses contact with the floor) Patient moves without compensation | 9 | Patient is instructed to lift pelvis from bed or table at the unaffected side (by shortening the unaffected side and lengthening | Patient demonstrates appropriate shortening/lengthening | |
| 1 Starting position Patient is instructed to rotate upper trunk 6 times (every shoulder should be moved forward 3 times), first side that moves must be hemiplegic side, head should be fixated in starting position 2 Repeat item 1 within 6 seconds Rotation is asymmetrical If score = 0, then item 2 scores 0 2 Repeat item 1 within 6 seconds Rotation is asymmetrical Rotation is asymmetrical Rotation is symmetrical 0 | 10 | Repeat item 9 | extremities, (2) pushing off with the ipsilateral foot (heel loses contact with the floor) Patient moves without compensation | □ 1 |
| Rotation is symmetrical | 1 | Starting position Patient is instructed to rotate upper trunk 6 times (every shoulder should be moved forward 3 times), first side that moves must be | Rotation is asymmetrical<br>Rotation is symmetrical | □ 1 |
| Patient is instructed to rotate lower trunk 6 times (every knee should be moved forward 3 times), first side that moves must be hemiplegic side, upper trunk should be fixated in starting position 4 Repeat item 3 within 6 seconds Rotation is asymmetrical If score = 0, then item 4 scores 0 Rotation is asymmetrical Rotation is asymmetrical Rotation is asymmetrical If score = 0, then item 4 scores 0 Rotation is asymmetrical If score = 0, then item 4 scores 0 Rotation is asymmetrical If score = 0, then item 4 scores 0 | 2 | Repeat item 1 within 6 seconds | | |
| Rotation is symmetrical 1 Total co-ordination /6 | 3 | Patient is instructed to rotate lower trunk 6 times (every knee should be moved forward 3 times), first side that moves must be | Rotation is asymmetrical<br>Rotation is symmetrical | |
| Total Trunk Impairment Scale /23 | 4 | Repeat item 3 within 6 seconds | Rotation is symmetrical | □ 1 |
| | | | Total Trunk Impairment Scale | /23 |



Maintaining Posture SUBTOTAL \_\_\_

## 1-3 PASS

## Maintaining a Posture

Give the subject instructions for each item as written below. When scoring the item, record the lowest response category that applies for each item.

| 1. Sitting Without Support |
|---|
| Examiner: Have the subject sit on a bench/mat without back support and with feet flat on the floor. |
| (3) Can sit for 5 minutes without support |
| (2) Can sit for more than 10 seconds without support |
| (1) Can sit with slight support (for example, by 1 hand) |
| (0) Cannot sit |
| 2. Standing With Support |
| Examiner: Have the subject stand, providing support as needed. Evaluate only the ability to stand with or without support. Do not consider the quality of the stance. |
| (3) Can stand with support of only 1 hand |
| (2) Can stand with moderate support of 1 person |
| (1) Can stand with strong support of 2 people |
| (0) Cannot stand, even with support |
| 3. Standing Without Support |
| Examiner: Have the subject stand without support. Evaluate only the ability to stand with or without support. Do not consider the quality of the stance. |
| (3) Can stand without support for more than 1 minute and simultaneously perform arm<br>movements at about shoulder level |
| (2) Can stand without support for 1 minute or stands slightly asymmetrically |
| (1) Can stand without support for 10 seconds or leans heavily on 1 leg |
| (0) Cannot stand without support |
| 4. Standing on Nonparetic Leg |
| Examiner: Have the subject stand on the nonparetic leg. Evaluate only the ability to bear weight entirely on the nonparetic leg. Do not consider how the subject accomplishes the task. |
| (3) Can stand on nonparetic leg for more than 10 seconds |
| (2) Can stand on nonparetic leg for more than 5 seconds |
| (1) Can stand on nonparetic leg for a few seconds |
| (0) Cannot stand on nonparetic leg |
| 5. Standing on Paretic Leg |
| Examiner: Have the subject stand on the paretic leg. Evaluate only the ability to bear weight entirely on the paretic leg. Do not consider how the subject accomplishes the task. |
| (3) Can stand on paretic leg for more than 10 seconds |
| (2) Can stand on paretic leg for more than 5 seconds |
| (1) Can stand on paretic leg for a few seconds |
| (0) Cannot stand on paretic leg |

#### Safety evaluation criteria and evaluation methods

Before starting the experiments, the health and physical condition of the subjects are assessed, and within 24 hours after the experiment, and signs of physical abnormalities are monitored.

## Data analysis and statistical methods

To determine the sample size, the G \* Power V.3.1 was utilized (Franz Paul, Kiel, Germany) (Faul F et al., 2007) incorporating an effect size of 0.44,  $\alpha$  < 0.05, power = 0.80, requiring total sample size of 12 participants (Dos Santos et al., 2019).

- 1. Statistical analysis was performed with IBM SPSS (version 28.0.1.1 (14)). Data were tested for normality using the Kolmogorov-Smirnov test. Kinematic data did not significantly deviate from a normal
- 2. distribution (P > 0.05). The Chi-square test was used to assess the sex distribution of the participants. The independent t-test and Mann-Whitney U test, as a nonparametric test, were employed to compare the two groups concerning specific demographic and clinical characteristics.

In the event of an unforeseen emergency, the participant's condition will be assessed, and immediate contact

## Predicted side effects and precautions with corresponding measures

will be made with emergency medical personnel for necessary actions. Subsequently, a prompt report will be submitted to the Institutional Review Board (IRB)

## Criteria for discontinuation and dropout

- 1. Inability to independently perform the action of sitting and extending the paralyzed arm
- 2. Feeling of dizziness

## Risks and benefits to research participants

- Prior to the start of the experiment, participants will receive a comprehensive explanation of the entire experimental procedure and the potential risks involved through an informed consent document. They will proceed with the experiment after understanding and acknowledging these risks.
- In the event of an emergency during the experiment, participants will be provided with non-monetary measures to seek medical examination and treatment from a qualified healthcare institution, even after the conclusion of the experiment.

#### References



Alt Murphy, M., Murphy, S., Persson, H. C., Bergström, U.-B., & Stibrant Sunnerhagen, K. (2018). Analysis Using 3D Motion Capture of Drinking Task in People With and Without Upper-extremity Impairments. J. Vis. Exp, 133, 57228. https://doi.org/10.3791/57228

Butcher, S. J., Craven, B. R., Chilibeck, P. D., Spink, K. S., Grona, S. L., & Sprigings, E. J. (2007). The effect of trunk stability training on vertical takeoff velocity. Journal of Orthopaedic and Sports Physical Therapy, 37(5), 223–231. https://doi.org/10.2519/JOSPT.2007.2331

Che-Nan, H., & Rambely, A. S. (2022). Kinematic Analysis of Daily Activity of Touching Lateral Shoulder for Normal Subjects. Applied Sciences (Switzerland), 12(4). https://doi.org/10.3390/APP12042069

Dean (1997) 'Task-related training improves performance of seated reaching tasks after stroke. A randomized controlled trial.', Stroke, 28(4), pp. 722–8. doi:info:doi/.

Murphy, M. A., Sunnerhagen, K. S., Johnels, B., & Willén, C. (2006). Three-dimensional kinematic motion analysis of a daily activity drinking from a glass: a pilot study. Journal of Neuroengineering and Rehabilitation, 3. https://doi.org/10.1186/1743-0003-3-18

Murphy, M. A., Willén, C., & Sunnerhagen, K. S. (2011). Kinematic variables quantifying upper-extremity performance after stroke during reaching and drinking from a glass. Neurorehabilitation and Neural Repair, 25(1), 71–80. https://doi.org/10.1177/1545968310370748

Norton, K. I. (2019). Standards for Anthropometry Assessment. In Kinanthropometry and Exercise Physiology (pp. 68–137). Routledge. https://doi.org/10.4324/9781315385662-4

Thrane, G., Thrane, G., Sunnerhagen, K. S., & Murphy, M. A. (2020). Upper limb kinematics during the first year after stroke: The stroke arm longitudinal study at the University of Gothenburg (SALGOT). Journal of NeuroEngineering and Rehabilitation, 17(1). https://doi.org/10.1186/s12984-020-00705-2

Winter, D. A. (2009). Biomechanics and motor control of human movement. Wiley.

Yang, S. H., Chung, E. J., Lee, J., Lee, S. H., & Lee, B. H. (2021). The effect of trunk stability training based on visual feedback on trunk stability, balance, and upper limb function in stroke patients: A randomized control trial. Healthcare (Switzerland), 9(5). https://doi.org/10.3390/HEALTHCARE9050532

Yang, S.-H., Chung, E.-J., Lee, J., Lee, S.-H., Lee, B.-H., & The, B. (2021). The Effect of Trunk Stability Training Based on Visual Feedback on Trunk Stability, Balance, and Upper Limb Function in Stroke Patients: A Randomized Control Trial Effect of Trunk Stability Training Based on Visual Feedback on Trunk



Stability, Balance, and Upper Limb Function in Stroke Patients: A Randomized Control Trial. Healthcare. <a href="https://doi.org/10.3390/healthcare9050532">https://doi.org/10.3390/healthcare9050532</a>